CLINICAL TRIAL: NCT01369017
Title: A Study of the Effect of Interleukin-1 Receptor Antagonist on Inhalation of 20,000 EU Clinical Center Reference Endotoxin in Normal Volunteers
Brief Title: Effect of Interleukin-1 Receptor Antagonist on Inhalation of 20,000 EU Clinical Ctr Reference Endotoxin in Normal Volunteers
Acronym: Kintox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michelle Hernandez, MD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Michelle Hernandez, MD, Assistant Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11-1026; 1U19AI077437-03 (NIH)
Record Dates: First submitted 2011-06-03; First posted 2011-06-08 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Control Subjects
Keywords: healthy volunteer; endotoxin
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anakinra (Active Comparator): All subjects will undergo 2 CCRE challenges. Each subject will be given either anakinra or placebo prior to CCRE challenge
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Normal saline injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Active treatment will consist of 2 doses of 1 mg/kg up to 100 mg of anakinra SQ injection.
  Arms: Anakinra
Drug: Placebo — Injection of NS
  Arms: Placebo

SUMMARY:
The investigators want to see if healthy people who are given 2 doses of a medication called anakinra, which is used to treat moderate to severe rheumatoid arthritis, (RA) and then exposed to a form of air pollution, called Endotoxin, have less inflammation with the medication. Endotoxin is believed to be one of the causes of asthma attacks.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* age 18-50 years

Exclusion Criteria:

* asthma
* pregnant women
* smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
blockade of IL-1 β will suppress neutrophil response to challenge with 20,000 EU CCRE | 6 hours after inhalation of CCRE
  The primary endpoints for this study will be a) safety assessments of anakinra with CCRE inhalation and b) the post CCRE challenge percentage of neutrophils (%PMN) in airway sputum during the anakinra treatment period compared to the placebo treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — UNC CH SOM
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States